CLINICAL TRIAL: NCT03951012
Title: Use Peripheral Blood Proteomics to Predict the Treatment Response and Toxicities in NSCLC Immunotherapy
Status: Terminated | Type: Observational
Why Stopped: low enrollment and remaining oncologist workload
Sponsor: Muhammad Furqan (Other)
Collaborators: Biodesix, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Muhammad Furqan, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201710764
Record Dates: First submitted 2019-04-17; First posted 2019-05-15 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants will be approached during their regular clinic visits and asked if an extra tube of blood may be collected prior to the treatment. If consent is not obtained before this visit, a participant will be asked later in the same day. The amount of blood collected will be 2 teaspoons (10mL).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood draw — Participants will be approached during their regular clinic visits and asked if an extra tube of blood may be collected prior to the treatment. If consent is not obtained before this visit, a participant will be asked later in the same day. The amount of blood collected will be 2 teaspoons (10mL).

SUMMARY:
Peripheral blood contains enormous quantity of biological information that can improve our patient care. Investigators plan to use proteomics from serum to study its value in predicting the therapeutic response and toxicities of immunotherapy in non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
An extra tube of blood for research will be collected from consented subjects prior to the initiation of anti-PD-1/L1 based immunotherapy, either single agent or in combination with chemotherapy. The blood will be coded, processed and sent for analysis. Results of analysis will be correlated with clinical data to see whether serum proteomics can be a good therapeutic predictor for future studies and treatments of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Non Small Cell Lung Cancer (NSCLC) patients who were previously untreated receiving anti-PD1 or anti-PD-L1 therapies, either single agent or in combination with chemotherapy.
* NSCLC patients who were treated with one previous line of therapy (not containing IO) and now receiving anti-PD1 or anti-PD-L1 therapies, either single agent or in combination with chemotherapy.

Exclusion Criteria:

* Patients not capable of making medical decisions
* Any patients who do not meet the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are current patients at Holden Comprehensive Cancer Center undergoing immunotherapy for Non Small Cell Lung Cancer (NSLC) prior to first chemotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Treatment response | Time of study enrollment up to one year
  Treatment response will be measured every 2-3 months using iRECIST criteria.
Treatment toxicities | Time of study enrollment up to one year
  The treatment toxicities will be recorded using CTCAE version 5.0
Correlate peripheral blood proteomics data with patients' clinical information | Time of study enrollment up to one year
  An extra tube of peripheral blood (~10ml) will be collected prior to the treatment. This blood specimen will be spun down and the serum collected and aliquoted. ~1ml serum will be shipped to Biodesix Inc. for the analysis of blood proteomics using matrix-assisted laser/desorption ionization (MALDI) mass spectrometry. We will correlate proteomics data with patients clinical information including treatment response, toxicities, tumor mutation/PD-L1 status, etc. to determine if peripheral blood protemoics can predict therapeutic response.

CONTACTS AND LOCATIONS:
Overall Officials: Taher Abu Hejleh, MBBS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ascierto PA, Capone M, Grimaldi AM, Mallardo D, Simeone E, Madonna G, Roder H, Meyer K, Asmellash S, Oliveira C, Roder J, Grigorieva J. Proteomic test for anti-PD-1 checkpoint blockade treatment of metastatic melanoma with and without BRAF mutations. J Immunother Cancer. 2019 Mar 29;7(1):91. doi: 10.1186/s40425-019-0569-1. PMID 30925943
- [Background] Quandt D, Dieter Zucht H, Amann A, Wulf-Goldenberg A, Borrebaeck C, Cannarile M, Lambrechts D, Oberacher H, Garrett J, Nayak T, Kazinski M, Massie C, Schwarzenbach H, Maio M, Prins R, Wendik B, Hockett R, Enderle D, Noerholm M, Hendriks H, Zwierzina H, Seliger B. Implementing liquid biopsies into clinical decision making for cancer immunotherapy. Oncotarget. 2017 Jul 18;8(29):48507-48520. doi: 10.18632/oncotarget.17397. PMID 28501851